CLINICAL TRIAL: NCT04404283
Title: A Randomized, Double-blind, Placebo-Controlled, Active-Comparator, Multicenter, Phase 3 Study of Brentuximab Vedotin or Placebo in Combination With Lenalidomide and Rituximab in Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Brentuximab Vedotin Plus Lenalidomide and Rituximab for the Treatment of Relapsed/Refractory DLBCL
Acronym: ECHELON-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGN35-031; C5691003 (Other: Alias Study Number); 2023-503384-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Seattle Genetics
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Brentuximab Vedotin; Rituximab; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Brentuximab vedotin + lenalidomide + rituximab
  Interventions: Drug: Brentuximab vedotin; Drug: Rituximab; Drug: Lenalidomide
- Control Arm (Active Comparator): Placebo + lenalidomide + rituximab
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Other: Placebo

INTERVENTIONS:
Drug: Brentuximab vedotin — 1.2 mg/kg administered into the vein (IV; intravenously) infusion every 3 weeks
  Arms: Experimental Arm
Drug: Rituximab — 375 mg/m^2 administered via intravenous infusion on Cycle 1 Day 1. 1400 mg injected under the skin (subcutaneous) permitted every 3 weeks from Cycle 2 Day 1 through end of treatment.
Drug: Lenalidomide — 20 mg given by mouth (orally) daily
Other: Placebo — Administered via intravenous infusion every 3 weeks
  Arms: Control Arm

SUMMARY:
Participants in this study will have diffuse large B-cell lymphoma (DLBCL) that has come back or not gotten better with treatment. The trial will study whether brentuximab vedotin plus two drugs works better to treat this type of cancer than the two drugs alone.

Participants will be randomly assigned to get either brentuximab vedotin or placebo. The placebo will look like brentuximab vedotin, but has no medicine in it. Since the study is "blinded," participants and their doctors will not know whether a participant gets brentuximab vedotin or placebo. All participants in the study will get rituximab and lenalidomide. These are drugs that can be used to treat DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Participants with relapsed or refractory diffuse and transformed large B-cell lymphoma (R/R DLBCL). DLBCL and cell of origin (GCB versus non-GCB) will be histologically determined by local pathology assessment for the purposes of study eligibility and stratification.
* Participants must have R/R disease following 2 or more lines of prior systemic therapy.

  * For participants with transformed DLBCL, at least the last systemic therapy used must have been for DLBCL
* Participants must be HSCT or CAR-T ineligible according to the investigator and must meet at least one of the following criteria:

  1. One or more co-morbidities, including cardiac, pulmonary, renal or hepatic dysfunction that in the opinion of the Investigator make the participant medically unfit to received HSCT or CAR-T therapy
  2. Active disease following induction and salvage chemotherapy
  3. Inadequate stem cell mobilization (for HSCT)
  4. Relapse following prior HSCT or CAR-T
  5. Unable to receive CAR-T therapy due to financial, geographic, insurance, or manufacturing issues
* Participants must have tumor tissue submitted to the central pathology lab. The tumor tissue submitted should be from the most recent biopsy that contains DLBCL.
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
* Participants must have fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET) and bidimensional measurable disease of at least 1.5 cm by computed tomography (CT), as assessed by the site radiologist within 28 days of Day 1.

Exclusion Criteria:

* History of another malignancy within 2 years before the first dose of study drug or any evidence of residual disease from a previously diagnosed malignancy
* History of progressive multifocal leukoencephalopathy (PML)
* Active cerebral/meningeal disease related to the underlying malignancy. Participants with a history of cerebral/meningeal disease related to the underlying malignancy are allowed if prior CNS disease has been effectively treated and without progression for at least 3 months.
* Any uncontrolled Grade 3 or higher (per NCI CTCAE version 5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study drug. Routine antimicrobial prophylaxis is permitted
* Chemotherapy, radiotherapy, biologics, and/or other antitumor treatment with immunotherapy that is not completed 3 weeks prior to first dose of study drug, unless underlying disease has progressed on treatment
* Previous treatment with brentuximab vedotin or lenalidomide.

  * Previous treatment with other vedotin-based ADCs is permitted if the last dose is at least 6 months prior to Day 1.
* Current therapy with immunosuppressive medications (including steroids), other systemic anti-neoplastic, or investigational agents

  a) Prednisone (or equivalent) ≤10 mg/day may be used for non-lymphomatous purposes
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class III-IV within 6 months prior to the first dose of study drugs
* Congestive heart failure, Class III or IV, by the NYHA criteria
* Grade 2 or higher peripheral sensory or motor neuropathy at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Approximately 2 years
  OS is defined as the time from the date of randomization to date of death due to any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Approximately 1 year
  PFS is defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. Assessment of PD will be performed by the investigator based on the Lugano Criteria for Response Assessment (Cheson 2014)
Objective response rate (ORR) | Approximately 1 year
  Proportion of participants with best response of complete response (CR) or partial response (PR) according to investigator assessment per the Lugano Criteria for Response Assessment (Cheson 2014).
Complete response (CR) rate | Approximately 1 year
  Proportion of participants with best response of CR according to investigator assessment per the Lugano Criteria for Response Assessment (Cheson 2014)
Duration of response (DOR) | Approximately 1 year
  Time from start of the first documentation of objective tumor response (CR or PR) to the first documentation of tumor progression by investigator assessment per the Lugano Criteria for Response Assessment (Cheson 2014) or death due to any cause, whichever occurs first.
Incidence of adverse events | Approximately 1 year
  Any untoward medical occurrence in a clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
OS in CD30+ participants | Approximately 2 years
  Time from the date of randomization to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (163):
- United States (45):
  - Central Alabama Research, Birmingham, Alabama
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Stuart, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Florida Cancer Specialists, Vero Beach, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - MidAmerica Division, Inc. c/o Menorah Medical Center, Overland Park, Kansas
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - IP ADDRESS: Brigitte Harris Cancer Pavilion (BHCP), Detroit, Michigan
  - Karmanos Cancer Institute Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Siteman Cancer Center - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - MidAmerica Division, Inc. c/o Centerpoint Medical Center, Independence, Missouri
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - Barnes Jewish-Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Siteman Cancer Center - North County, St Louis, Missouri
  - Oncology_Hematology Care Clinical Trials,LLC, Cincinnati, Ohio
  - University of Cincinnati Medical Center IDS Pharmacy, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oncology_Hematology Care Clinical Trials,LLC, Fairfield, Ohio
  - West Chester Hospital, West Chester, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Roper St. Francis Healthcare, Mt. Pleasant, South Carolina
  - Roper St. Francis Healthcare, North Charleston, South Carolina
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center, Irving, Texas
  - University of Virginia Cancer Center., Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
- Australia (10):
  - Central Coast Local Health District, Gosford Hospital, Gosford, New South Wales
  - Central Coast Local Health District Wyong Hospital, Hamlyn Terrace, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Breakthrough Haematology Hollywood Specialist Centre, Nedlands, Western Australia
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - Bellberry Limited, Eastwood
  - Ramsay National Research Unit and Research Governance Office, Greenslopes
  - Tasmania Health and Medical HREC, Hobart
  - Hollywood Haematology, Nedlands
- Belgium (6):
  - CHU UCL Namur-, Yvoir, Namur
  - ZNA Middelheim, Antwerp
  - ZNA Cadix, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Chu Helora, Haine-Saint-Paul
- Canada (7):
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - CISSS de la Monteregie-Centre, Greenfield Park, Quebec
  - Centre Integre Universitaire de la Santé et de Services Sociaux de l'Est-de-l'ile-de-Montreal,, Montreal, Quebec
  - Centre Integre Universitaire De Sante et de Services Sociaux Du Nord-de-I'ile-de-Montreal, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Lekarna Fakultni nemocnice Hradec Kralove, Hradec Králové
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Clinical Trial Unit 2081, Copenhagen
  - Nuklearmedicin, Copenhagen
  - Zealand University Hospital Roskilde, Roskilde
- France (23):
  - Centre de Lutte Contre le Cancer (CLCC) - Institut Bergonie, Bordeaux, Other
  - Centre Hospitalier(CH) de Perpignan, Perpignan, Other
  - Hôpital Lyon Sud, Pierre-Bénite, Other
  - CHU Angers - Hotel Dieu Nord, Service des Maladies du Sang, Angers
  - Centre de Lutte Contre le Cancer (CLCC) - lnstitut Bergonie Pharmacie, Bordeaux
  - Centre Hospitalier Metropole Savoie, Chambéry
  - Centre Hospitalier Sud Francilien (CHSF), Corbeil-Essonnes
  - CHU Grenoble Alpes, Grenoble
  - Centre Hospitalier Le Mans, Le Mans
  - Pharmacie a Usage lnterieur CHU de LIMOGES, Limoges
  - Service d'Hematologie Clinique, Limoges
  - CHR Metz-Thionville Hopital Mercy, Metz
  - Centre Hospitalier Universitaire Nantes-Hotel Dieu, Service d'Hematologie, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Saint-Antoine -, Paris
  - Service Pharmacie Essais Cliniques Centre Hospitalier (CH) de Perpignan, Perpignan
  - Service d'Hematologie clinique et Therapie cellulaire CHU Bordeaux Hopital Haut-Leveque, Pessac
  - Pharmacie Hopital Haut-Leveque Unite des Essais Cliniques, Pessac
  - Centre Henri Becquerel, Rouen
  - Service de Radiologie ,Centre Henri Becquerel, Rouen
  - CHRU Hopital de Tours, Tours
  - CHRU de Nancy - Hopitaux de Brabois, Service Hematologie et Medecine interne, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy Département d'Innovations Thérapeutiques et d'Essais Précoces (DITEP), Villejuif
- ICON Laboratory Services, Leopardstown, Other, Ireland
- Italy (5):
  - IRCCS Istituto Tumori Giovanni Paolo II U.O. Ematologia, Bari, Apulia
  - Azienda Ospedaliera "Cardinale Giovanni Panico", U.O.C. Ematologia e Trapianti Midollo Osseo, Tricase, Lecce
  - Istituto Europeo di Oncologia, Milan, MI
  - Azienda Ospedaliero-Universitaria di Bologna - IRCCS, Bologna, Other
  - Ospedale Maggiore ASUGI, Trieste
- Poland (4):
  - Voxel S.A., Krakow
  - Pratia MCM Krakow, Krakow
  - Zaklad Rentgena i Usg - Wyrobek Sp. z o.o. sp. k, Krakow
  - Nasz Lekarz Osrodek Badan Klinicznych, Torun
- South Korea (13):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - The Catholic University of Korea, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital., Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital Yonsei University Health System, Seoul
  - SoonChunHyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul Saint Mary's Hospital, Seoul
- Spain (23):
  - Hospital San Pedro de Alcantara, Cáceres, Extremadura
  - Hospital Universitario QuironSalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Costa del Sol, Marbella, Malaga
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona, Other
  - Hospital Universitario de Badajoz, Badajoz
  - Assaigs Clfnics-Servei de Farmacia, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Quiron, Barcelona
  - Cetir, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital La Milagrosa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - FUNDAClON GENERAL UNIVERSIDAD DE MALAGA (FGUMA), Málaga
  - Hospital Rey Juan Carlos, Móstoles
  - Hospital Universitario QuironSalud Madrid, Pozuelo de Alarcon (madrid)
  - Centro de Diagnostico y Resonancia Magnetica, Salamanca
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Switzerland (5):
  - Univ. Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Winterthur, Medizinische Onkologie, Winterthur, Canton of Zurich
  - Universitatsspital Zurich, Zurich, Other
  - Universitatsspital Basel, Basel
  - Kantonsapotheke Zurich, Schlieren
- Taiwan (9):
  - National Taiwan University Hospital Clinical Trial Pharmacy, Taipei, R.o.c
  - National Taiwan University Hospital, Taipei, R.o.c
  - Chang Gung Medical Foundation, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - Chi Mei Medical Center, Liouying, Tainan
  - Pharmacy Department, Taipei Veterans General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, WEST Midlands
  - St Bartholomew's hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, Sandwich

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Bartlett NL, Hahn U, Kim WS, Fleury I, Laribi K, Bergua JM, Bouabdallah K, Forward N, Bijou F, MacDonald D, Portell CA, Ghesquieres H, Nowakowski G, Yasenchak CA, Patterson M, Ho L, Rustia E, Fanale M, Jie F, Kim JA. Brentuximab Vedotin Combination for Relapsed Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2025 Mar 20;43(9):1061-1072. doi: 10.1200/JCO-24-02242. Epub 2025 Jan 7. PMID 39772655
- [Derived] Ward JP, Berrien-Elliott MM, Gomez F, Luo J, Becker-Hapak M, Cashen AF, Wagner-Johnston ND, Maddocks K, Mosior M, Foster M, Krysiak K, Schmidt A, Skidmore ZL, Desai S, Watkins MP, Fischer A, Griffith M, Griffith OL, Fehniger TA, Bartlett NL. Phase 1/dose expansion trial of brentuximab vedotin and lenalidomide in relapsed or refractory diffuse large B-cell lymphoma. Blood. 2022 Mar 31;139(13):1999-2010. doi: 10.1182/blood.2021011894. PMID 34780623
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGN35-031